CLINICAL TRIAL: NCT03849625
Title: Characteristics of Patients Diagnosed With NSAID Sensitivity in Thailand
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Jettanong Klaewsongkram, MD., Assoc. Prof. Jettanong Klaewsongkram, MD., Chulalongkorn University
Other Study IDs: Chula-ARC 002/13
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Aspirin Sensitivity; Aspirin-exacerbated Respiratory Disease; Aspirin-Induced Angioedema-Urticaria; Aspirin Allergy; NSAID-Induced Asthma; NSAID-Induced Angioedema-Urticaria; NSAID-Induced Anaphylactoid Reaction; Aspirin-Induced Anaphylactoid Reaction
MeSH Terms: conditions — Asthma, Aspirin-Induced | interventions — Aspirin; Anti-Inflammatory Agents, Non-Steroidal; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSAID sensitivity: Patients diagnosed with an immediate reaction to aspirin/NSAIDs/or paracetamol
  Interventions: Drug: aspirin, NSAIDs, paracetamol

INTERVENTIONS:
Drug: aspirin, NSAIDs, paracetamol — Perform skin test and/or provocation test with aspirin, paracetmol, or suspected NSAIDs in questionable cases

SUMMARY:
Study clinical characteristics and phenotypes of patients diagnosed with NSAID sensitivity in Thailand

ELIGIBILITY:
Inclusion Criteria:

* Thai patients with a history of an immediate reaction to aspirin/paracetamol, or NSAIDs visiting King Chulalongkorn memorial Hospital

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at least 15 years of age with a history of an immediate reaction to aspirin/paracetamol, or NSAIDs
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Results of skin test/provocation test | 4 years
  Positive, negative, or equivocal

SECONDARY OUTCOMES:
Phenotypes of allergic reactions | 4 years
Urine leukotriene E4 | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klaewsongkram J, Buranapraditkun S, Mongkolpathumrat P, Palapinyo S, Chantaphakul H. Clinical Characteristics, Urinary Leukotriene E4 Levels, and Aspirin Desensitization Results in Patients With NSAID-Induced Blended Reactions. Allergy Asthma Immunol Res. 2021 Mar;13(2):229-244. doi: 10.4168/aair.2021.13.2.229. PMID 33474858